CLINICAL TRIAL: NCT03819413
Title: Clinical Patterns of Neuromyelitis Optica Spectrum Disorders in Assiut University Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, doaa mokhtar mahmoud, Principal Investigator, Assiut University
Other Study IDs: NMOSD In Assiut University
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Neuromyelitis Optica Spectrum Disorder; prevalence; anti-AQP4; anti-MOG
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum aquaporin 4 antibody (AQP-4-Ab) — All patients suspected to have NMOSD according to the recent diagnostic criteria will be examined for serum aquaporin 4 antibody (AQP-4-Ab) and serum myelin oligodendrocyte glycoprotein antibody (anti-MOG)
Diagnostic Test: serum MOG antibody (anti-MOG) — All patients suspected to have NMOSD according to the recent diagnostic criteria will be examined for serum myelin oligodendrocyte glycoprotein antibody (anti-MOG) if they tested negative for serum aquaporin 4 antibody (AQP-4-Ab)
Diagnostic Test: MRI brain, spine and orbit — All patients suspected to have NMOSD according to the recent diagnostic criteria will have MRI brain, spine and orbit with Gadolinium

SUMMARY:
Neuromyelitis Optica Spectrum Disorders (NMOSD) are a group of inflammatory demyelinating disorders of the central nervous system. Although NMOSD occurs much more commonly in nations with a predominately non-Caucasian population, NMOSD are underestimated in Egypt and frequently misdiagnosed as multiple sclerosis (MS). In this study, by investigating serum anti-aquaporin (AQP) 4 and anti-MOG antibody of patients suspected to have NMOSD attending the Neurology and Psychiatry department of Assiut University Hospital, investigators aim to determine the relative frequency, clinical and radiological characteristics of NMOSD in upper Egypt community and compare it with other populations of different races.

DETAILED DESCRIPTION:
Neuromyelitis Optica Spectrum Disorders (NMOSD) are a group of inflammatory demyelinating disorders of the central nervous system characterized by episodes of immune-mediated demyelination and axonal damage mainly involving optic nerves and spinal cord. The discovery of a disease-specific serum NMO-immunoglobulin G (IgG) antibody that selectively binds aquaporin-4 (AQP4) has not only distinguish NMO from MS but also enabled an appreciation for the wide spectrum of this disorder. Another autoantibody is the Myelin oligodendrocyte glycoprotein (MOGIgG) antibody that has been increasingly reported in a variety of central nervous system neuroinflammatory conditions including patients with phenotypes typical for NMOSD. Overall, NMO occurs much more commonly in nations with a predominately non-Caucasian population,and estimated to be as high as 10 per 100,000. Differentiation of MS from NMOSD is critically important because disease modifying treatment for MS, are inefficacious in or may aggravate NMOSD. However, in Africa and Middle East, publications and studies are rare and most often focus on isolated cases that clearly do not reflect the epidemiological reality in this area. Investigators believe that detailed assessment of serum AQP4 antibody as well as anti-MOG antibody in Egyptian patients with suspected NMOSD or those with idiopathic inflammatory demyelinating central nervous system diseases (IIDCD) other than typical MS would be beneficial and Eventually will help to avoid unnecessary investigations and treatments, recurrent and prolonged hospital course, significant morbidity, and even death.

ELIGIBILITY:
Inclusion Criteria:

* All cases that fulfill the international 2015 consensus criteria of NMOSD
* Any episode suggestive of idiopathic inflammatory demyelinating central nervous system disease including

  * longitudinally extensive transverse myelitis (LETM) or optic neuritis (ON) plus Cerebral or Brainstem syndrome (LETM or ON PLUS)
  * optic neuritis (ON)
  * longitudinally extensive transverse myelitis (LETM),
  * Transverse myelitis with non-extensive lesion (NETM)
  * Acute encephalomyelitis (ADEM).
* Atypical MS cases (atypical clinical presentation, course, radiological findings or atypical response to treatment)
* Age: all patients of both sexes and all age groups will be included.

Exclusion Criteria:

* Inclusion criteria for suspected NMOSD were not met
* An alternate diagnosis became apparent
* if no serum sample was supplied
* Subject declined to provide written informed consent.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients suspected to have NMOSD according to the recent diagnostic criteria attending or referred to Neurology and Psychiatry department of Assiut University hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
the percentage of increase in NMOSD diagnostic rates by screening for serum anti-AQP4 and anti-MOG antibodies | one year period
  To assess the role of screening for Serum anti-AQP4 and anti-MOG antibodies in patients with idiopathic inflammatory central nervous system demyelinating disorders on diagnostic rates of NMOSD

SECONDARY OUTCOMES:
percentage of patients were misdiagnosed as MS after screening for serum anti-AQP4 and anti-MOG antibodies | one year period
  To measure the role of Serum anti-AQP4 and anti-MOG antibodies to differentiate suspicious cases from MS
the percentage of increase of anti-MOG associated diseases after screening for serum anti-MOG antibodies | one year period
  To assess the impact of screening for serum anti-MOG antibodies on diagnostic rates of anti-MOG associated diseases

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Abo Elfotoh, prof, Study Director — Assuit university hospital
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weinshenker BG, Wingerchuk DM. Neuromyelitis Spectrum Disorders. Mayo Clin Proc. 2017 Apr;92(4):663-679. doi: 10.1016/j.mayocp.2016.12.014. PMID 28385199
- [Background] Pandit L, Asgari N, Apiwattanakul M, Palace J, Paul F, Leite MI, Kleiter I, Chitnis T; GJCF International Clinical Consortium & Biorepository for Neuromyelitis Optica. Demographic and clinical features of neuromyelitis optica: A review. Mult Scler. 2015 Jun;21(7):845-53. doi: 10.1177/1352458515572406. Epub 2015 Apr 28. PMID 25921037
- [Background] Lennon VA, Wingerchuk DM, Kryzer TJ, Pittock SJ, Lucchinetti CF, Fujihara K, Nakashima I, Weinshenker BG. A serum autoantibody marker of neuromyelitis optica: distinction from multiple sclerosis. Lancet. 2004 Dec 11-17;364(9451):2106-12. doi: 10.1016/S0140-6736(04)17551-X. PMID 15589308
- [Background] Di Pauli F, Reindl M, Berger T. New clinical implications of anti-myelin oligodendrocyte glycoprotein antibodies in children with CNS demyelinating diseases. Mult Scler Relat Disord. 2018 May;22:35-37. doi: 10.1016/j.msard.2018.02.023. Epub 2018 Feb 22. PMID 29524760
- [Background] Kim SM, Kim SJ, Lee HJ, Kuroda H, Palace J, Fujihara K. Differential diagnosis of neuromyelitis optica spectrum disorders. Ther Adv Neurol Disord. 2017 Jul;10(7):265-289. doi: 10.1177/1756285617709723. Epub 2017 May 24. PMID 28670343
- [Background] Holroyd KB, Aziz F, Szolics M, Alsaadi T, Levy M, Schiess N. Prevalence and characteristics of transverse myelitis and neuromyelitis optica spectrum disorders in the United Arab Emirates: A multicenter, retrospective study. Clin Exp Neuroimmunol. 2018 Aug;9(3):155-161. doi: 10.1111/cen3.12458. Epub 2018 May 7. PMID 30090123
- [Background] Jarius S, Paul F, Aktas O, Asgari N, Dale RC, de Seze J, Franciotta D, Fujihara K, Jacob A, Kim HJ, Kleiter I, Kumpfel T, Levy M, Palace J, Ruprecht K, Saiz A, Trebst C, Weinshenker BG, Wildemann B. MOG encephalomyelitis: international recommendations on diagnosis and antibody testing. J Neuroinflammation. 2018 May 3;15(1):134. doi: 10.1186/s12974-018-1144-2. PMID 29724224